CLINICAL TRIAL: NCT04523792
Title: Virginia Opioid Treatment-Emergency Department
Acronym: VOT-ED
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funder has not approved protocol
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Indivior, PLC. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20020289
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Opioid Use Disorder
Keywords: Opioid use disorder; Opioid withdrawal; Emergency department; Treatment-seeking; Opioid agonist treatment; Sublocade
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies | interventions — Sublocade

STUDY DESIGN:
Intervention Model Description: The study is designed to examine feasibility of SUBLOCADE on outpatient treatment engagement compared to historical and concurrent control groups.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Opioid withdrawal patients (Experimental): Subjects with opioid use disorder seeking treatment and/or experiencing symptoms of opioid withdrawal receive acute administration of SUBOXONE sublingual film followed by SUBLOCADE administration in the 1) ED, 2) Clinical Decision Unit or 3) Inpatient unit combined with 6 months of treatment with SUBLOCADE in the outpatient treatment clinic.
  Interventions: Drug: SUBLOCADE

INTERVENTIONS:
Drug: SUBLOCADE — SUBLOCADE (buprenorphine extended-release) injection is a colorless to amber sterile solution for SC injection designed to deliver buprenorphine at doses of 100 mg or 300 mg at a controlled rate over a one-month period.

SUMMARY:
The current study seeks to test the feasibility of an alternative treatment for patients with opioid use disorder who present to the emergency department seeking treatment or with opioid withdrawal, which includes FDA approved long-acting medication for opioid misuse (SUBLOCADE) and rapid transfer of care to outpatient substance abuse treatment.

DETAILED DESCRIPTION:
This proof of concept study will provide feasibility data on whether rapid initiation of SUBLOCADE® (buprenorphine extended-release) injection for subcutaneous use CIII in the ED, Clinical Decision Unit, or inpatient unit and after administration of a test dose of SUBOXONE® (buprenorphine and naloxone) sublingual film, for sublingual or buccal use CIII among treatment-seeking adults with moderate or severe OUD increases subsequent outpatient treatment engagement as compared to a historical control cohort and concurrent controls who decline treatment participation. The study will also assess whether rapid initiation of SUBLOCADE® reduces subsequent ED visits for any reason. As a exploratory aim we will examine whether rapid initiation of Sublocade in this patient group reduces opioid overdose events compared to historical controls and patients who decline Sublocade.

ELIGIBILITY:
Inclusion criteria:

1. Signed the informed consent form (ICF) and have the ability to comply with the requirements and restrictions listed therein.
2. Age: ≥ 18 years at time of executing the ICF.
3. Currently meets DSM-5 criteria for moderate to severe OUD.
4. Is clinically stable (respiratory rate [RR] ≥ 12, pulse oximetry > 95%, Glasgow Coma Scale [GCS] score of 15) and suitable for the trial in investigator's or designee's judgement.
5. Agrees not to take any buprenorphine products other than those administered during the current study throughout participation in the study.
6. Negative urine pregnancy test for females.
7. Vital signs (BP, HR, temperature) considered within normal limits or non-clinically significant elevation, as assessed by treating physician.
8. Provide a urine drug screen positive for illicit opioids, excluding methadone.
9. Have a COWS score ≥ 8.
10. Is seeking medication-assisted treatment for OUD.

Exclusion Criteria:

1. Current diagnosis, other than OUD, requiring chronic opioid treatment.
2. Active suicidal ideation in opinion of the Investigator or designee.
3. Female subject that is lactating, pregnant or planning to become pregnant during their participation in the study.
4. Uncontrolled intercurrent illness including, but not limited to, psychiatric illness that would limit compliance with study requirements or compromise the ability of the subject to provide written informed consent.
5. Known allergy or hypersensitivity to SUBOXONE or SUBLOCADE.
6. Any condition that, in the opinion of the Investigator would interfere with interpretation of subject safety or study results.
7. Currently receiving methadone, depot naltrexone, or Probuphine for OUD or received those treatments for OUD within 30 days prior to consent.
8. Current or concurrent treatment with an investigational agent.
9. Current or concurrent enrollment in another clinical study, or observational study that includes MAT.
10. Treatment for OUD required by court order.
11. Current or pending incarceration/legal action that could affect participation or compliance in the study.
12. Subjects who are unable, in the opinion of the Investigator, to comply fully with the study requirements.
13. Less than 48-72 hours since last use of long acting opioids (i.e., methadone), by self-report.
14. Current intoxication with benzodiazepines or alcohol.
15. Meet current DSM-5 diagnosis for severe Benzodiazepine or Alcohol Use Disorder or endorse benzodiazepine or alcohol withdrawal symptoms.
16. Current illicit opioid users who endorse regular use of long acting opioids (i.e., methadone).
17. Total bilirubin ≥ 1.5x the upper limit of normal (ULN), alanine aminotransferase (ALT) ≥3xULN, aspartate aminotransferase (AST) ≥ 3xULN, serum creatinine > 2xULN, international normalized ratio (INR) >1.5xULN. If these results are unable to be obtained prior to enrolling the subject, the investigator can make an initial determination about eligibility based on LFTs collected in the past 6 months from the subject's medical record.
18. Patients with a history of Long QT Syndrome or an immediate family member with this condition or those taking Class lA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide) or Class Ill antiarrhythmic medications (e.g., sotalol, amiodarone) or other medications that prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment engagement - 1 month | 1 month
  Treatment engagement as measured by percentage of participants who attend an outpatient clinic visit within 1 month of first injection.

SECONDARY OUTCOMES:
Treatment engagement - 3 and 6 months | 3 and 6 months
  Treatment engagement as measured by percentage of participants who continue to attend outpatient clinic visits with SUBLOCADE injections (buprenorphine treatment) at 3 and 6 months.
Number of repeat ED visits | 6 months
  Number of repeat ED visits for any reason will be measured from electronic medical records and self-reported data.

OTHER OUTCOMES:
Healthcare resource utilization | 6 months
  Healthcare resource utilization (measured by number of outpatient clinic and emergency department visits, and number of inpatient admissions) as compared to the concurrent and historical control groups.
Opioid craving | 6 months
  Opioid craving in subjects as measured by Craving Visual Analog Scale (VAS), a 3-item scale in which individuals rate their cravings for opioids on a scale from 0 (NOT AT ALL) to 10 (EXTREMELY).
Number of participants with a urine drug screen negative for illicit opioids. | 6 months
  Illicit opioid use as measured by urine drug screen (UDS) results.
Impulse control | 6 months
  Time to decision in delay discounting task
Opioid cravings | 6 months
  Brief opioid demand task
Number of non-fatal or fatal opioid-related overdoses | 6 months
  Data on the number of opioid overdoses will be measured from electronic medical records and/or state death registries.
Treatment effectiveness: Treatment Effectiveness Assessment (TEA) | 6 months
  Treatment effectiveness as measured by Treatment Effectiveness Assessment (TEA), which measures on 4 domains (substance use, health, lifestyle, community involvement). Responses on each item range from 1 ("not better at all") to 10 ("very much better") with items summed for a total score of 4-40, and higher scores reflecting greater self-report of treatment effectiveness.
Medication satisfaction: Medication Satisfaction Questionnaire (MSQ) | 6 months
  Measured by the Medication Satisfaction Questionnaire (MSQ), a single item that asks participants to rate how satisfied they are with their current opioid dependence medication on a scale from 1 ("extremely dissatisfied") to 7 ("extremely satisfied"). Higher scores reflect greater satisfaction with the medication.
Employment, presentism and absenteeism | 6 months
  Assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP), which measures the effects of opioid use disorder on the ability to work and perform regular activities among participants. Items evaluate hours of work completed and hours of work missed in the past 7 days and ask participants to rate the impact on their work productivity and regular activities in the past 7 days on a scale of 0 ("problem had no effect on my work/regular activities") to 10 ("problem completely prevented me from working/regular activities"), with higher scores reflecting greater severity and worse outcomes on the measure.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University